CLINICAL TRIAL: NCT03494374
Title: The Effect of Orthosis and Exercise in Pes Planus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ju Seok Ryu (Other)
Responsible Party: Sponsor-Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-1701/377-303
Record Dates: First submitted 2018-04-02; First posted 2018-04-11 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pes Planus
Keywords: pes planus; UCBL; exercise
MeSH Terms: conditions — Flatfoot; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Annual evaluation after applying UCBL and exercise treatment. Cohort study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Treatment with UCBL and exercise therapy
  Interventions: Device: UCBL orthosis

INTERVENTIONS:
Device: UCBL orthosis — toe walking exercise
  Other Names: Exercise

SUMMARY:
There is no definite evidence for the conservative treatment of pes planus. We want to verify the combination efficacy of orthosis and toe walking exercise for the treatment of pes planus.

DETAILED DESCRIPTION:
Observation cohort study

We prescribe UCBL orthosis and teach toe walking exercise. And we will check standing foot radiography (AP/Lateral) annually. And we will compare the changes of talometatarsal angle and calcaneal pitch angle.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with pes planus
* Calcaneal pitch angle < 15 degree

Exclusion Criteria:

* peripheral neuropathy
* infection
* rheumatoid arthritis
* operation history

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-12-29 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
TM angle | through study completion, an average of 1 year
  Talometatarsal angle

SECONDARY OUTCOMES:
CP angle | through study completion, an average of 1 year
  Calcaneal pitch angle

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes